CLINICAL TRIAL: NCT03818724
Title: Treatment Success With the CoolLoop Cryoablation System - Post-Market Surveillance
Brief Title: Treatment Success With the CoolLoop Cryoablation System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: afreeze GmbH (Other)
Collaborators: Raffeiner GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CooL-TreatS
Record Dates: First submitted 2019-01-21; First posted 2019-01-28 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases
Keywords: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Cryoablation; Cryosurgery
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CoolLoop® cryoablation system: Cryoablation for treatment of atrial fibrillation using the CoolLoop® cryoablation system
  Interventions: Device: CoolLoop® cryoablation system

INTERVENTIONS:
Device: CoolLoop® cryoablation system — Cryoablation of Atrial Fibrillation using the CoolLoop® Cryoablation System

SUMMARY:
This clinical study evaluates the safety and efficacy of the treatment with the CoolLoop® cryoablation System (sclerotherapy of muscle tissue of the heart by freezing) in patients with atrial fibrillation (permanent atrial fibrillation excepted) over a follow-up period of 36 months.

A further aim of this study is to evaluate the average duration of procedure and fluoroscopy times.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* atrial fibrillation: permanent AF excepted
* ECG documented AF within the last 6 months
* patients planned for an ablation procedure and suitable and planned for treatment with the CoolLoop® cryoablation system
* signed and dated informed consent documented by the patient, indicating that the patient has been informed of all the pertinent aspects of the trial prior to study enrollment (patient has received a copy of the ICF)

Exclusion Criteria:

* indication that the vascular system is not accessible through the left or right groin.
* indication that a transseptal puncture cannot be performed.
* any previous ablation or surgery due to AF.
* important comorbidities such as cardiovascular events within six months of enrollment or high-risk surgical patients.
* pregnant women at the time of the cryoablation procedure.
* any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the Informed Consent Form.
* participation in interventional trials for cardiovascular devices or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have to be planned and be suitable for an ablation procedure. The decision to treat the patients with the CoolLoop® cryoablation System has already been made in advance by the Investigator. Informed consent has to be obtained before the ablation procedure.
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events | 36 months follow-up period
  Safety is measured by the percentage of participants with serious adverse events (SAEs) up to 36 months post-ablation
Freedom from atrial fibrillation (efficacy) at 36 months post-ablation | 36 months follow-up period
  Efficacy is measured by the percentage of AF (atrial fibrillation) free patients at 36 months post-ablation

SECONDARY OUTCOMES:
Freedom from atrial fibrillation (efficacy) at 12 and 24 months post-ablation | 12 and 24 months post-ablation
  Efficacy is measured by the percentage of AF (atrial fibrillation) free patients at 12 and 24 months post-ablation
Acute procedure success | 36 months follow-up period
  Acute efficacy of isolation of each of the pulmonary veins defined as the percentage of diagnostic mapping catheter electrode pairs within the pulmonary vein without any detectable pulmonary vein signal in case of redo procedure
Total procedure time | Estimated timeframe up to 4 hours
  Total procedure time defined from introduction of the sheath until removal of the sheath
CoolLoop procedure time | Estimated timeframe up to 2 hours
  CoolLoop procedure time defined from introduction of the CoolLoop cryoablation catheter into the left atrium until removal from the left atrium after Termination of the last cryo-application with the CoolLoop cryoablation catheter
Total fluoroscopy time | Estimated time frame up to 1 hour
  Total fluoroscopy time defined from introduction of the sheath until removal of the sheath
CoolLoop fluoroscopy time | Estimated timeframe up to 30 minutes
  CoolLoop fluoroscopy time defined from introduction of the CoolLoop cryoablation catheter into the left atrium until removal from the left atrium after termination of the last cryo-application with the CoolLoop cryoablation catheter
Cumulative cryoablation time | Estimated timeframe up to 1 hour
  Cumulative cryoablation time is displayed as "total freeze time" by the cryoconsole at the end of the procedure
Adverse Events (AEs) of special interest | 36 months follow-up period
  Recording of AEs of Special interest and patient reported cardiac arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kaiser, PhD, Study Director — afreeze GmbH; Florian Hintringer, MD, Principal Investigator — Medical University Innsbruck
Locations (2):
- Medical University Innsbruck, Innsbruck, Tirol/Austria, Austria
- Marienhaus Klinikum St. Elisabeth Neuwied, Neuwied, Germany/Rheinland-Pfalz, Germany